CLINICAL TRIAL: NCT01305265
Title: Post-operative Sore Throat as Determines by Endotracheal Tube Inflation Technique
Brief Title: Post-operative Sore Throat as Determined by Endotracheal Tube Inflation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: weottp
Record Dates: First submitted 2011-02-24; First posted 2011-02-28 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Post Operative Sore Throat; Dysphagia; Hoarseness
Keywords: sore throat; dysphagia; hoarseness; post operative; endotracheal intubation
MeSH Terms: conditions — Deglutition Disorders; Hoarseness; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): Endotracheal tube will be adjusted to 22-26 cm H20 pressure immediately post intubation using a cuff manometer
  Interventions: Device: cuff manometer
- control (No Intervention): endotracheal tube cuff will be inflated using standard technique

INTERVENTIONS:
Device: cuff manometer — endotracheal tube cuff will be inflated to 22-26 cm H20 using cuff manometer
  Arms: intervention

SUMMARY:
The purpose of this study is to test whether the incidence of sore throat and other tracheal co-morbidities such as dysphagia and hoarseness can be lessened by use of a cuff manometer at the beginning of surgery to inflate to the proper pressure compared to the standard technique.

The investigators hypothesis is that inflation of the endotracheal balloon using a cuff manometer immediately after intubation will reduce the incidence of sore throat and other tracheal co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for general anesthesia requiring endotracheal intubation with planned duration of at least 2 hours
* ASA I-3

Exclusion Criteria:

* Planned prolonged intubation
* Planned postoperative ICU admission
* Non English speaking
* Mentally impaired
* Existing tracheal stoma
* Nasogastric tube in place preoperative
* Thyroid / intra-oral surgery
* Previous general anesthesia within the last 2 weeks
* Use of steroids within one week before surgery (IV,inhaled, oral)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Endotracheal tube cuff will be inflated using the inflate&palpate technique
- Intervention Group: Endotracheal tube cuff will be inflated using the inflate & palpate technique. The cuff pressure will be adjusted to 22-26cmH2O within 15min after intubation by trained study staff.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 71 | 70
Completed | 69 | 64
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Endotracheal tube cuff inflated using the inflate & palpate technique
- Intervention Group: Endotracheal tube cuff inflated using the inflate & palpate technique. The cuff pressure then was adjusted to 22-26cmH2O within 15min after endotracheal intubation by trained study staff.
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 69 | 64 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (15.8) | 50.3 (13.8) | 51.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 37 | 30 | 67
Region of Enrollment [Number; unit: participants]
  United States | 69 | 64 | 133

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Tracheopharyngeal Symptoms
Time Frame: within 2 hours after extubation
Measure: Number; unit: participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 69 | 64
participants | 53 | 49

ADVERSE EVENTS:
Arm/Group | Control Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/64
Other Adverse Events (participants affected / at risk) | 0/69 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes